CLINICAL TRIAL: NCT06448806
Title: Epigenetic Signature of Advance Glycation End Products (AGE) and Skin Autofluorescence As a Risk Predictor in Metabolically Healthy and Unhealthy Obese Adults
Brief Title: Mobile Health (M-health) Intervention to Reduce the Epigenetic Signature in Metabolic Syndrome (MetS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sadia Fatima, Associate Professor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Mhealth-Epigen
Record Dates: First submitted 2024-05-21; First posted 2024-06-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifestyle modification through m-health (Other): Individuals recruited will be followed for a year and offered lifestyle intervention
  Interventions: Other: mobile health lifestyle intervention

INTERVENTIONS:
Other: mobile health lifestyle intervention — You will be asked to record all dietary and physical activity log for 12 months on an application. Mobile sms reminders will be sent to you on regular basis. At day 0, at 6th and 12 months you will be asked to provide 3 ml of blood for the methylation and advance glycation level testing and your weight and body fat percentage will be measured. During this period you will have to follow the lifestyle and diet chart provided to you by the researchers.

SUMMARY:
The goal of this interventional study is to learn about the improvement in body composition effects of lifestyle intervention in subjects with metabolic syndrome. The main question it aims to answer is:

Does life style intervention lower body fat% and gene methylation levels in subjects with metabolic syndrome? Participants will answer survey questions and get blood and body composition testing done at day 0, at 6 months and 12 months. Keep a diary of their food and activity and the number of times they use mobile health application.

DETAILED DESCRIPTION:
This is same as above.

ELIGIBILITY:
Inclusion Criteria:

1. Less than 5 kg body weight fluctuation in the 6 months prior to recruitment.
2. Ideal body weight for height falling according to the South Asian Criteria as per WHO recommended i.e. Body Mass Index (BMI) of 18.5 to 22.9 kg/m2 (normal-weight) and above 23kg/m2 (overweight/ obese).
3. Any one of the following characteristics "according to the modified National Cholesterol Education Program (NCEP) ATPIII guidelines i) waist circumference ii) hyper triglyceridemia (triglycerides ≥150 mg/dl) or low High density lipoprotein (HDL) cholesterol (HDL cholesterol ≤40 mg/dl for men and ≤50 mg/dl for women iii) elevated blood pressure (systolic blood pressure ≥130 mmHg and/or diastolic blood pressure ≥85 mmHg or current use of antihypertensive drugs) iv) impaired fasting glucose (fasting plasma glucose ≥100mg/dl) v) waist circumference (90 cm in men and 80 cm in women)".
4. Have access to a smart phone/mobile and not using the fitness application

Exclusion Criteria:

1. Age <18 or above 65 year
2. Pregnant women
3. Individuals with other comorbidities such as cancers, hepatic and/or renal impairment, or on hormonal supplements and/or anti-inflammatory drugs etc.
4. Unfit for blood testing or no smart phone available

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Weight in kilograms, height in meter (will be combined to report BMI in kg/m^2) | one year
  A weighing scale will be used for this and values recorded on a questionnaire
Advance glycation end product (U/mL) from serum | one year
  This serum biomarker level will be assessed by Enzyme linked immunosorbent assay (ELISA) at the laboratory. Values will be recorded as Units per milliliter on a questionnaire.
Body fat percentage | 1 year
  Body composition will be measured by Bioelectrical impedance matching (BIA) and computerized topography (CT) scans. The reports will be shared with the participants and values will be recorded on a questionnaire.

SECONDARY OUTCOMES:
Methylation level of genes | 1 year
  From the blood samples collected, DNA will be used to measure the methylation level of genes of interest such as Leptin, Ghrelin, fat mass obesity, chemerin etc. These molecular biology testing of this physiological parameter will be conducted in the laboratory and results will be recorded on a questionnaire.
Meal quality and calorie count | 1 year
  Participants will be asked to make a meal diary and write all their food intake and physical activity on a mobile app. They will share their monthly progress with the investigator via WhatsApp (m-health) .

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Fatima, PhD, Principal Investigator — Aga Khan University
Locations (1):
- DBBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No